CLINICAL TRIAL: NCT03340844
Title: Role of Circulating Tumor Cells (CTC´s) Spread During Pancreaticoduodenectomy in Metastasis and Survival Rates in Patients With Pancreatic and Periampullary Tumors
Brief Title: Role of CTC´s Spread During Pancreaticoduodenectomy in Patients With Pancreatic and Periampullary Tumors
Acronym: CETUPANC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CETUPANC
Record Dates: First submitted 2017-10-16; First posted 2017-11-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Tumor; Periampullary Carcinoma Resectable; Circulating Tumor Cells; Metastasis
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (1:1) to 2 study groups according to duodenopancreatectomy surgical approach: "No-Touch group" (NT) or "Artery First group" (SMA) in patients with pancreatic and periampullary tumors, to evaluated circulating tumor cells (CTCs) levels during the surgery. Sample size = 86
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Touch (NT) (Experimental): Pancreatic and Periampullary Tumors resection by no-touch technique
  Interventions: Procedure: No Touch (NT)
- Superior Mesenteric Artery First (SMA) (Active Comparator): Pancreatic and Periampullary Tumors resection by superior Mesenteric Artery First technique
  Interventions: Procedure: Superior Mesenteric Artery First (SMA)

INTERVENTIONS:
Procedure: No Touch (NT) — Tumor resection by No-touch technique: dissection of hepatic hilum, dissection of superior mesenteric vein (SMV) in caudal aspect of pancreas, section of antrum, pancreatic neck section. Section-ligation of veins of duodenopancreatectomy part of SMV and portal. Then Kocher-uncrossing maneuver of the jejunal loop and final section of the retro-portal (back of the portal vein) blade.
  Arms: No Touch (NT)
Procedure: Superior Mesenteric Artery First (SMA) — Tumor resection by SMA technique: Kocher maneuver extends to the left renal vein (LRV). Dissection above the LRV of the SMA (refer to vessel-loop). Then, SMA will be identified on the caudal side of the pancreas (mesenterial root) and progressive dissection until its origin in the aorta artery (previously referenced with vessel loop).
  Arms: Superior Mesenteric Artery First (SMA)

SUMMARY:
This multicentre, prospective and randomized study aims(1:1) to compare the rate of recurrence, metastasis and survival according to the levels of intraoperative circulating tumor cells (CTCs) during cephalic duodenopancreatectomy in patients with pancreatic and periampullary tumors.

DETAILED DESCRIPTION:
Cephalic duodenopancreatectomy is the technique indicated for patients with pancreatic head carcinoma and periampullar tumors.

There are different technical variants, it is not standardized what is the best option in relation to local recurrence, metastasis and survival.

In the study, patients will be randomized into two study groups with pancreatic and periampullary tumors undergoing cephalic pancreatectomy (NT) vs initial approach by superior mesenteric artery (SMA).

The measurement of circulating tumor cells (CTCs) allows to assess the degree of cellular dissemination due to surgical manipulation.CTCs will be evaluated during surgery (nº CTCs / mL blood). To do this, a maximum of 4 blood samples from the portal vein will be performed, in each study group according to the following scheme:

* NT group: basal (at the beginning of surgery), portal vein pancreatic detachment, postresection (NT2) and before closure (NT3).
* SMA group: basal (at the beginning of surgery), after Kocher maneuver and SMA dissection, postresection, before closure.

Subsequently, the quantified levels of CTCs will be correlated with the occurrence of local tumor recurrence, metastasis development and patient patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years, with adenocarcinomas of the pancreas and potentially resectable periampullary tumors by cephalic duodenopancreatectomy or total duodenopancreatectomy indicated intraoperatively for technical reasons, who voluntarily agree to participate in the study and sign informed consent

Exclusion Criteria:

1. Patients in whom liver metastases or peritoneal carcinomatosis are detected during surgery.
2. Patients with neuroendocrine pancreatic tumors or cystic tumors.
3. Patients in whom tumor resection is not finally achieved because it shows intraoperatively that the tumor is locally advanced and unresectable.
4. Patients with macroscopic residual tumor (R2).
5. High-risk patients with severe pathology (ASA IV) according to the American Association of Anesthesiologists.
6. Patients receiving neoadjuvant therapy
7. Patients in whom the intraoperative pathological anatomy indicates borders of pancreatic resection affected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Circulating tumor cells (CTC´s) | During the surgery: at the beginning of surgery, immediately after disconnecting the pancreas from the portal vein, just at the moment the pancreatic resection ends and before the skin closed
  Change in the concentration of circulating tumor cells (CTCs) levels (nº CTCs/ mL blood) during the surgery, 4 blood samples will be taken from the portal vein
Local tumor recurrence | From the day of surgery to 3 years of follow-up
  Presence (YES or NO) compatible images of local tumor recurrence Valid imaging tests of presence or absence can be checked by: computerized tomography (CT) or magnetic resonance (NMR)
Metastasis | From the day of surgery to 3 years of follow-up
  Presence (YES or NO) compatible images of metastasis
Patient survival | From the day of surgery to 3 years of follow-up
  Death (YES OR NO): number of patients dying during study

SECONDARY OUTCOMES:
Morbidity | From the day of surgery up to 6 weeks of follow-up
  The complications evaluation and their severity will be based on the classification of Dindo-Clavien and the definitions of the International Study Group of Pancreatic Surgery (ISGPS).
  * Pancreatic fistula: Presence (yes or no) and degree (A, B, C)
  * Delayed gastric emptying: Presence (yes or no) and degree (A, B, C)
  * Hemorrhage: Presence (yes or no) and degree (A, B, C)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Padillo Ruiz, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Yes. Anonymized data for individual participant data (IPD) is planned to be shared with all participants within 6 months of data completion
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within 6 months after database closure and analysis.

REFERENCES:
- [Background] Matsuno S, Egawa S, Fukuyama S, Motoi F, Sunamura M, Isaji S, Imaizumi T, Okada S, Kato H, Suda K, Nakao A, Hiraoka T, Hosotani R, Takeda K. Pancreatic Cancer Registry in Japan: 20 years of experience. Pancreas. 2004 Apr;28(3):219-30. doi: 10.1097/00006676-200404000-00002. PMID 15084961
- [Background] Kutomi G, Mizuguchi T, Satomi F, Maeda H, Shima H, Kimura Y, Hirata K. Current status of the prognostic molecular biomarkers in breast cancer: A systematic review. Oncol Lett. 2017 Mar;13(3):1491-1498. doi: 10.3892/ol.2017.5609. Epub 2017 Jan 17. PMID 28454281
- [Background] Jamieson NB, Foulis AK, Oien KA, Going JJ, Glen P, Dickson EJ, Imrie CW, McKay CJ, Carter R. Positive mobilization margins alone do not influence survival following pancreatico-duodenectomy for pancreatic ductal adenocarcinoma. Ann Surg. 2010 Jun;251(6):1003-10. doi: 10.1097/SLA.0b013e3181d77369. PMID 20485150
- [Background] Alamo JM, Marin LM, Suarez G, Bernal C, Serrano J, Barrera L, Gomez MA, Muntane J, Padillo FJ. Improving outcomes in pancreatic cancer: key points in perioperative management. World J Gastroenterol. 2014 Oct 21;20(39):14237-45. doi: 10.3748/wjg.v20.i39.14237. PMID 25339810
- [Background] Sabater L, Calvete J, Aparisi L, Canovas R, Munoz E, Anon R, Rosello S, Rodriguez E, Camps B, Alfonso R, Sala C, Sastre J, Cervantes A, Lledo S. [Pancreatic and periampullary tumors: morbidity, mortality, functional results and long-term survival]. Cir Esp. 2009 Sep;86(3):159-66. doi: 10.1016/j.ciresp.2009.03.014. Epub 2009 Jul 18. Spanish. PMID 19616203
- [Background] Verbeke CS, Menon KV. Redefining resection margin status in pancreatic cancer. HPB (Oxford). 2009 Jun;11(4):282-9. doi: 10.1111/j.1477-2574.2009.00055.x. PMID 19718354
- [Background] Earl J, Garcia-Nieto S, Martinez-Avila JC, Montans J, Sanjuanbenito A, Rodriguez-Garrote M, Lisa E, Mendia E, Lobo E, Malats N, Carrato A, Guillen-Ponce C. Circulating tumor cells (Ctc) and kras mutant circulating free Dna (cfdna) detection in peripheral blood as biomarkers in patients diagnosed with exocrine pancreatic cancer. BMC Cancer. 2015 Oct 24;15:797. doi: 10.1186/s12885-015-1779-7. PMID 26498594
- [Background] Connor AA, McNamara K, Al-Sukhni E, Diskin J, Chan D, Ash C, Lowes LE, Allan AL, Zogopoulos G, Moulton CA, Gallinger S. Central, But Not Peripheral, Circulating Tumor Cells are Prognostic in Patients Undergoing Resection of Colorectal Cancer Liver Metastases. Ann Surg Oncol. 2016 Jul;23(7):2168-75. doi: 10.1245/s10434-015-5038-6. Epub 2015 Dec 29. PMID 26714949
- [Background] Poruk KE, Valero V 3rd, Saunders T, Blackford AL, Griffin JF, Poling J, Hruban RH, Anders RA, Herman J, Zheng L, Rasheed ZA, Laheru DA, Ahuja N, Weiss MJ, Cameron JL, Goggins M, Iacobuzio-Donahue CA, Wood LD, Wolfgang CL. Circulating Tumor Cell Phenotype Predicts Recurrence and Survival in Pancreatic Adenocarcinoma. Ann Surg. 2016 Dec;264(6):1073-1081. doi: 10.1097/SLA.0000000000001600. PMID 26756760
- [Background] BARNES JP. Physiologic resection of the right colon. Surg Gynecol Obstet. 1952 Jun;94(6):722-6. No abstract available. PMID 14931182
- [Background] Hirota M, Kanemitsu K, Takamori H, Chikamoto A, Tanaka H, Sugita H, Sand J, Nordback I, Baba H. Pancreatoduodenectomy using a no-touch isolation technique. Am J Surg. 2010 May;199(5):e65-8. doi: 10.1016/j.amjsurg.2008.06.035. Epub 2008 Dec 18. PMID 19095210
- [Background] Hirota M, Ogawa M. No-touch pancreatectomy for invasive ductal carcinoma of the pancreas. JOP. 2014 May 27;15(3):243-9. doi: 10.6092/1590-8577/2502. PMID 24865535
- [Background] Kobayashi S, Asano T, Ochiai T. A proposal of no-touch isolation technique in pancreatoduodenectomy for periampullary carcinomas. Hepatogastroenterology. 2001 Mar-Apr;48(38):372-4. PMID 11379311
- [Background] Gall TM, Jacob J, Frampton AE, Krell J, Kyriakides C, Castellano L, Stebbing J, Jiao LR. Reduced dissemination of circulating tumor cells with no-touch isolation surgical technique in patients with pancreatic cancer. JAMA Surg. 2014 May;149(5):482-5. doi: 10.1001/jamasurg.2013.3643. PMID 24599353
- [Background] Pessaux P, Marzano E, Rosso E. A plea for the artery-first dissection during pancreaticoduodenectomy. J Am Coll Surg. 2010 Jul;211(1):142-3. doi: 10.1016/j.jamcollsurg.2010.03.026. No abstract available. PMID 20610264
- [Background] Weitz J, Rahbari N, Koch M, Buchler MW. The "artery first" approach for resection of pancreatic head cancer. J Am Coll Surg. 2010 Feb;210(2):e1-4. doi: 10.1016/j.jamcollsurg.2009.10.019. Epub 2009 Dec 3. No abstract available. PMID 20113929
- [Background] Sanjay P, Takaori K, Govil S, Shrikhande SV, Windsor JA. 'Artery-first' approaches to pancreatoduodenectomy. Br J Surg. 2012 Aug;99(8):1027-35. doi: 10.1002/bjs.8763. Epub 2012 May 9. PMID 22569924
- [Background] Kuroki T, Eguchi S. No-touch isolation techniques for pancreatic cancer. Surg Today. 2017 Jan;47(1):8-13. doi: 10.1007/s00595-016-1317-5. Epub 2016 Mar 1. PMID 26931548
- [Derived] Padillo-Ruiz J, Fresno C, Suarez G, Blanco G, Munoz-Bellvis L, Justo I, Garcia-Domingo MI, Ausania F, Munoz-Forner E, Serrablo A, Martin E, Diez L, Cepeda C, Marin L, Alamo J, Bernal C, Pereira S, Calero F, Tinoco J, Paterna S, Cugat E, Fondevila C, Diego-Alonso E, Lopez-Guerra D, Gomez M, Denninghoff V, Sabater L. Effects of the superior mesenteric artery approach versus the no-touch approach during pancreatoduodenectomy on the mobilization of circulating tumour cells and clusters in pancreatic cancer (CETUPANC): randomized clinical trial. BJS Open. 2024 Oct 29;8(6):zrae123. doi: 10.1093/bjsopen/zrae123. PMID 39485887